CLINICAL TRIAL: NCT02868879
Title: Anatomical and Structural Connectivity in Schizophrenias
Brief Title: Anatomical and Structural Connectivity in Two Psychotic Phenotypes : Periodic Catatonia and Cataphasia
Status: Completed | Type: Observational
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Other Study IDs: 2898
Record Dates: First submitted 2016-08-05; First posted 2016-08-16 (Estimated); Last update posted 2019-10-21 (Actual); Status verified 2019-10

CONDITIONS: Schizophrenia; Catatonia
MeSH Terms: conditions — Schizophrenia; Catatonia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Schizophrenia
  Interventions: Other: Quantitative multiparametric and functional MRI
- Normal controls.
  Interventions: Other: Quantitative multiparametric and functional MRI

INTERVENTIONS:
Other: Quantitative multiparametric and functional MRI — Structural connectivity assessed in the cortex and the white matter using multimodal quantitative parametric imaging (R1, R2, R2*, DTI, susceptibility, macromolecular proton fraction, cortical thickness, VBM).
  Functional connectivity assessed using simple BOLD and combined ASL-BOLD sequences during multiple tasks including motor, language and working memory tasks.

SUMMARY:
The different subtypes of Schizophrenia might have a disordered connectivity as their final common pathways.

The investigators will use multimodal structural MRI to assess anatomical connectivity on the one side and its functional consequence on functional connectivity on the other side to assess two phenotypes of psychosis : periodic catatonia and cataphasia in comparison with control subjects.

The coherence between structural and functional anomalies will be especially studied.

ELIGIBILITY:
Inclusion criteria (controls):

* Aged from 18-65 Y
* Right handed

Additional inclusion criteria for patients:

* Schizophrenia according to the DSM5
* Either periodic catatonia or cataphasia according to the WKL classification
* Under stable medication regimen (> 1M)

Exclusion criteria:

* Current substance abuse
* Contraindication to MRI
* Past records susceptible to affect brain integrity
* Severe, unstable medical condition
* Pregnancy
* Patients deprived of their rights

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Schizophrenia patients (subdivided in periodic catatonia and cataphasia) and normal controls, both having the same procedure.
Sampling Method: Non-Probability Sample
Enrollment: 162 (Actual)
Dates: Start 2006-09-25 (Actual); Primary Completion 2019-09 (Actual); Study Completion 2019-09 (Actual)

PRIMARY OUTCOMES:
Changes in structural and functional connectivity according to the phenotype. Correlation between these changes | Subjects will be assessed only once.
  Statistical parametric mapping (SPM) will be applied on quantitative maps : rCBF (ml/100g/min), susceptibility (part per billion), R1, R2, R2* (all expressed in ms-1), fractional anisotropy (fraction), averaged diffusivity (μm²/sec), macromolecular proton fraction (percentage), cortical thickness (mm), VBM (probability of grey and white matter) and contrast maps (BOLD signal correlation with the anterior cingulate ROI).

SECONDARY OUTCOMES:
Changes in rCBF and cognition according to the phenotype. Correlation between the different changes and the symptomatic scales. | Subjects will be assessed only once.
  Symptomatic scales : PANSS, SANS, SAPS, Calgary, Bush and Francis catatonia scale, the psychological experimental test operationalized for cataphasia, Clinician-rated dimension of psychosis symptom severity questionnaire assessing handedness, anhedonia, vigilance, QoL, activity, handicap, ruminations, depression and personality.
  Cognitive tests : grammar tests, semantic priming, implicit memory, CPT, fNART, Mill-Hill (part B)

CONTACTS AND LOCATIONS:
Locations (1):
- Service de Psychiatrie, Hôpital Civil, Hôpitaux Universitaires de Strasbourg, Strasbourg, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Foucher JR, Zhang YF, Roser M, Lamy J, De Sousa PL, Weibel S, Vidailhet P, Mainberger O, Berna F. A double dissociation between two psychotic phenotypes: Periodic catatonia and cataphasia. Prog Neuropsychopharmacol Biol Psychiatry. 2018 Aug 30;86:363-369. doi: 10.1016/j.pnpbp.2018.03.008. Epub 2018 Mar 17. PMID 29559372